CLINICAL TRIAL: NCT07103018
Title: Phase 1, Dose-Escalation Study of KTX2001 (an NSD2 Inhibitor) Alone and in Combination With Darolutamide for Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Clinical Study of KTX-2001 in Subjects With Metastatic Castration-Resistant Prostate Cancer (STRIKE-001)
Acronym: STRIKE-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: K36 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: K36-MCRPC-001
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer Patients; Metastatic Castration-resistant Prostate Cancer, mCRPC; mCRPC; mCRPC (Metastatic Castration-resistant Prostate Cancer)
Keywords: mCRPC; Metastatic Castration-Resistant Prostate Cancer; castration-resistant prostate cancer; NSD2 inhibitor; efficacy; safety; pharmacokinetics; pharmacodynamics; Darolutamide; NUBEQA; Metastatic Disease; Neoplasms; prostatic Diseases; Prostatic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urogenital Diseases; Male Urogenital Diseases; Epigenetics
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Prostatic Diseases; Prostatic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urogenital Diseases; Male Urogenital Diseases | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation Monotherapy (Experimental): KTX-2001 orally
  Interventions: Drug: KTX-2001
- Part B: Dose Escalation Combination (Experimental): KTX-2001 orally Darolutamide (NUBEQA®) orally as 600 mg BID, total daily dose at 1200 mg
  Interventions: Drug: KTX-2001 + Darolutamide (NUBEQA®)

INTERVENTIONS:
Drug: KTX-2001 — Participants will receive escalating doses of KTX-2001 monotherapy
  Arms: Part A: Dose Escalation Monotherapy
Drug: KTX-2001 + Darolutamide (NUBEQA®) — Participants will receive escalating doses of KTX-2001, in combination with the oral androgen receptor (AR) pathway inhibitor (ARPI), darolutamide (NUBEQA®)
  Arms: Part B: Dose Escalation Combination

SUMMARY:
Study K36-MCRPC-001 is the first in human clinical trial testing KTX-2001 alone and with darolutamide in men with metastatic castration-resistant prostate cancer. The study aims to assess whether the drug is safe, increasing doses alone and in combination with darolutamide, whether it is effective in treating metastatic castration-resistant prostate cancer, and measuring how the drug(s) behaves in the body.

DETAILED DESCRIPTION:
Study K36-MCRPC-001 (also know as K36-STRIKE-001) is a multicenter, open-label Phase 1 study for participants with metastatic castration-resistant prostate cancer (mCRPC) to investigate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of KTX-2001 monotherapy and KTX-2001 in combination with darolutamide (NUBEQA®), and to establish a recommended Phase 2 dose(s) of KTX-2001 for future study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
3. Male participants with mCRPC as defined by PCWG3 criteria.
4. Metastatic disease documented using bone scan for bone metastases (PCWG3 criteria) or by computed tomography (CT) or magnetic resonance imaging (MRI) for soft-tissue metastases. Evidence of metastasis on prostate-specific membrane antigen positron emission tomography alone will not be sufficient for confirmation of metastatic disease.
5. Willingness to undergo a baseline and on-treatment biopsy of a metastatic site if safe and feasible. If tissue from a biopsy of a metastatic site (including bone) obtained within the previous 6 months (prior to treatment start) is available, this tissue may be used, and the baseline biopsy may be omitted.
6. Participants should have progressed on or after receiving an ARPI (eg, abiraterone, enzalutamide, darolutamide, or apalutamide).
7. Adequate renal function (creatinine clearance >50 mL/min by serum creatinine).
8. Adequate hepatic function (total bilirubin ≤1.5× ULN, total bilirubin <3× ULN for participants with documented Gilbert's syndrome, AST and ALT ≤2.5× ULN). In case of liver metastases, AST and ALT <5× ULN is allowed.
9. Adequate hematological function (neutrophils >1 × 109/L, platelet count >100 × 109/L, hemoglobin >9 g/dL) with no prior transfusions within 2 weeks.

Exclusion Criteria:

1. Presence of symptomatic or uncontrolled brain metastases unless adequately treated, not requiring steroids and stable for the last 28 calendar days before signing the ICF. Participants with leptomeningeal disease are excluded without exception.
2. Symptomatic or impending cord compression that has not been treated or stabilized.
3. Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction (such as coagulopathy or encephalopathy), or other reasons which, in the investigator's opinion, could compromise the participant's safety or interfere with or compromise the integrity of the study outcomes.
4. Presence of a drug-related toxicity from prior cancer therapy that has not resolved to Grade ≤1 (with the exception of alopecia and Grade 2 neuropathy) according to NCI-CTCAE Version 5.0.
5. Active, uncontrolled, bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness. In equivocal cases, participants with a negative viral load may be eligible. Eligibility criteria for HIV-positive participants currently on highly active antiretroviral therapy should be evaluated and discussed with the medical monitor and will be based on current and past CD4 and T cell counts, history (if any) of AIDS-defining conditions (eg, opportunistic infections), and status of HIV treatment. Participants with previously treated HBV and HCV with negative viral load are eligible.
6. A significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that, in the opinion of the investigator, would adversely affect participation in this study.

   1. QT interval corrected by Fridericia's formula >470 msec at screening.
   2. Unstable cardiovascular function defined as:
   3. Symptomatic ischemia, or
   4. Uncontrolled clinically significant conduction abnormalities (ie, ventricular tachycardia on antiarrhythmic agents are excluded; first-degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block are not excluded), or
   5. Congestive heart failure New York Heart Association Class ≥3, or
   6. Myocardial infarction within 3 months of the screening visit.
   7. Hypertension that cannot be controlled (persistent >150/90 mmHg despite optimal medical therapy).
7. Current use or anticipated need for food or drugs that are known strong CYP3A inducers or inhibitors, including their administration within 10 days or 5 half-lives of the CYP3A inhibitor, whichever is longer prior to first dose of study drug.
8. Treatment with anticancer therapies including radiotherapy or AR-targeted therapy/androgen biosynthesis inhibitor) within 2 weeks prior to initial study drug dose or within 4 weeks for systemic chemotherapy, radioligand therapy, or other systemic anticancer therapies.
9. Treatment with another investigational agent in the 4 weeks prior to the initial dose of study drug.
10. Major surgical procedures ≤28 days prior to the initial dose of study drug. Participants must have recovered from any of the effects of any major surgery. No waiting period is required following central venous access placement, biopsy collection, or minor surgeries as long as the investigator assesses the impact on study participation.
11. Initiation of hormonal agents with antitumor activity against prostate cancer including 5alpha reductase inhibitors, androgens (eg, testosterone), cytoproterone acetate, etc during study participation (from the time of consent to off-study); however, stable use of 5-alpha reductase inhibitors is permitted, if continuous use for ≥6 months.
12. Use of herbal products or alternative therapies that may decrease PSA levels or that may have hormonal anti-prostate cancer activity (eg, saw palmetto, PC-SPES, PC-HOPE, St. John's wort, selenium supplements, grape seed extract, etc) within 4 weeks of study drug initiation or plans to initiate treatment with these products/alternative therapies at any point during the study.

For Part B only (KTX-2001 + darolutamide): Current use or anticipated need for drugs that are known as combined P-glycoprotein (P-gp) and strong or moderate CYP3A4 inducers including their administration within 10 days or 5 half-lives of the combined Pgp/CYP3A4 inducer, whichever is longer prior to first dose of darolutamide.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with dose-limiting toxicities (DLTs) to determine the maximum tolerated dose (MTD) | 21 days

SECONDARY OUTCOMES:
Overall safety profile including adverse events | up to 1095 days
Recommended Phase 2 dose (RP2D) of KTX-2001 | up to 1095 days
Pharmacokinetic Parameters: Maximum Observed Plasma Concentration (Cmax) | up to 48 hours
  Characterize PK parameters of KTX-2001 when administered as a single agent or in combination with darolutamide

CONTACTS AND LOCATIONS:
Overall Officials: Jason Redman, MD, Study Director — K36 Therapeutics
Locations (13):
- United States (13):
  - University of California San Francisco, San Francisco, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Mayo Clinic, Rochester, Minnesota
  - START New York Long Island, LLC, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Carolina Urologic Research Center, the START Center for Cancer Research, Myrtle Beach, South Carolina
  - USA Clinical Trials, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided